CLINICAL TRIAL: NCT01561313
Title: A Multicenter, Randomized, Single-Blind Crossover Study of the Safety and Tolerability of Two Adalimumab Formulations in Adult Subjects With Rheumatoid Arthritis.
Brief Title: Crossover Study of Safety and Tolerability of Two Formulations of Adalimumab.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: M12-783; 2011-002275-41 (EudraCT Number)
Record Dates: First submitted 2012-03-21; First posted 2012-03-23 (Estimated); Results first posted 2014-02-20 (Estimated); Last update posted 2014-02-20 (Estimated); Status verified 2014-01

CONDITIONS: Rheumatoid Arthritis
Keywords: On label Humira users; Pain; Rheumatoid Arthritis,
MeSH Terms: conditions — Arthritis, Rheumatoid; Pain | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Current formulation adalimumab (Active Comparator): One dose with 40 mg of current formulation of adalimumab in a pre-filled syringe
  Interventions: Biological: Adalimumab
- New formulation of adalimumab (Experimental): One dose with 40 mg of new formulation of adalimumab in a pre-filled syringe
  Interventions: Biological: Adalimumab

INTERVENTIONS:
Biological: Adalimumab — Subcutaneously 40 mg every other week (EOW) or every week (EW) (as dosing requires)
  Other Names: Humira; ABT-D2E7

SUMMARY:
This study will compare injection site pain levels between current Humira® formulation versus a new formulation of Humira in patients with Rheumatoid Arthritis (RA), who are either currently on a stable dose (minimum six consecutive doses) of on-label Humira or biological naïve who will be prescribed on-label Humira as treatment for their Rheumatoid Arthritis. The study is being conducted in two countries, Belgium (3 sites) and the Czech Republic (3 sites).

DETAILED DESCRIPTION:
64 participants were randomized, 63 received at least one dose of the study drug, and 62 participants were analyzed for injection site-related pain. 63 participants were analyzed for other safety analyses. Two participants, who were randomized to the Current formulation adalimumab/New formulation of adalimumab arm of the study were excluded from the analysis of injection site-related pain. One participant received one dose of study drug and discontinued because of an adverse event, while the other discontinued before receiving any study drug.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject age 18 years or older, who requires Humira 40 mg SC every other week (eow) or every week (ew) for the treatment of rheumatoid arthritis, in accordance with the local Humira label.
* Subject must be a current, on-label user of Humira who rates his/her average Humira injection site related pain as at least 3 cm on a pain Visual Analogue Scale and has had at least 6 consecutive doses of Humira prior to Screening, or a biologic naïve subject who requires initiation of on-label treatment with Humira.
* Subject has diagnosis of rheumatoid arthritis (RA) as defined by the 1987 revised ACR classification criteria or the ACR/EULAR 2010 criteria,
* Female subjects are either not of childbearing potential, defined as postmenopausal for at least 1 year or surgically sterile (bilateral tubal ligation, bilateral oophorectomy and/or hysterectomy), or are practicing at least one method of birth control throughout the study and for at least 70 days after the last dose of study drug.
* All female subjects of childbearing potential must have a negative test for pregnancy on a serum sample at Screening and prior to study drug dosing on a urine sample obtained at Visit 1.

Exclusion Criteria:

* Subject has been treated with any investigational drug of a chemical or biologic nature within a minimum of 30 days or 5 half-lives (whichever is longer) of the drug prior to Visit 1.
* Any infection(s) requiring treatment with intravenous (IV) anti-infectives within 30 days prior to Visit 1 or oral anti-infectives within 14 days prior to Visit 1.
* Prior exposure to natalizumab (Tysabri®) or efalizumab (Raptiva®).
* Known hypersensitivity to adalimumab or its excipients.
* History of demyelinating disease (including myelitis) or neurologic symptoms suggestive of demyelinating disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2012-03; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Payne, PhD, Study Director — AbbVie
Locations (6):
- Belgium (3):
  - Site Reference ID/Investigator# 63357, Genk
  - Site Reference ID/Investigator# 63359, Ghent
  - Site Reference ID/Investigator# 63360, Ghent
- Czechia (3):
  - Site Reference ID/Investigator# 63363, Brno
  - Site Reference ID/Investigator# 63362, Prague
  - Site Reference ID/Investigator# 63361, Uherské Hradiště

REFERENCES:
- [Derived] Nash P, Vanhoof J, Hall S, Arulmani U, Tarzynski-Potempa R, Unnebrink K, Payne AN, Cividino A. Randomized Crossover Comparison of Injection Site Pain with 40 mg/0.4 or 0.8 mL Formulations of Adalimumab in Patients with Rheumatoid Arthritis. Rheumatol Ther. 2016 Dec;3(2):257-270. doi: 10.1007/s40744-016-0041-3. Epub 2016 Aug 18. PMID 27747583
- See also: This clinical study may be evaluating a usage that is not currently FDA-approved. Please see US prescribing information for approved uses. — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two participants, who were randomized to the Current formulation adalimumab/New formulation of adalimumab arm of the study, were excluded from the analysis of injection site-related pain. One participant received one dose of study drug and discontinued because of an adverse event, while the other discontinued before receiving any study drug.
Groups:
- Current Formulation Adalimumab/New Formulation of Adalimumab: First dose with 40 mg of current formulation of adalimumab in a pre-filled syringe and second dose with 40 mg of new formulation of adalimumab in a pre-filled syringe.
- New Formulation of Adalimumab/Current Formulation Adalimumab: First dose with 40 mg of new formulation of adalimumab in a pre-filled syringe and second dose with 40 mg of current formulation of adalimumab in a pre-filled syringe.
Period: Overall Study
Arm/Group | Current Formulation Adalimumab/New Formulation of Adalimumab | New Formulation of Adalimumab/Current Formulation Adalimumab
Started | 33 | 31
Completed | 31 | 31
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse event and withdrawal by subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: 63 participants received at least one dose of the study drug, and 62 participants were analyzed for injection site-related pain. 63 participants were analyzed for other safety analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | Current Formulation Adalimumab/New Formulation of Adalimumab | New Formulation of Adalimumab/Current Formulation Adalimumab | Total
Number analyzed (Participants) | 31 | 31 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.1 (12.57) | 58.6 (13.53) | 54.8 (13.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 21 | 42
  Male | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Mean Injection Site Pain on a Visual Analogue Scale (VAS)
Description: The primary response variable is participant's immediate pain of injection on a visual analogue scale (VAS) of 0 to 10 (cm), with 0 representing no pain and 10 representing the worst possible pain.
Time Frame: Immediately after injection
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Current Formulation Adalimumab | New Formulation of Adalimumab
Number analyzed (Participants) | 62 | 62
cm | 3.3 (2.11) | 1.6 (2.09)

2. Secondary Outcome: Mean Injection Site Pain on a Visual Analogue Scale (VAS)
Description: The secondary response variable is participant's pain of injection on a visual analogue scale (VAS) of 0 to 10 (cm) recorded 15 minutes after the injection, with 0 representing no pain and 10 representing the worst possible pain.
Time Frame: 15 minutes post injection
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Current Formulation Adalimumab | New Formulation of Adalimumab
Number analyzed (Participants) | 62 | 62
cm | 1.0 (1.52) | 0.9 (1.66)

3. Secondary Outcome: Percentage of Participants With no Hemorrhage/Petechiae in the Draize Scale
Description: Hemorrhage/petechiae (bleeding/spots of bleeding underneath the skin) was assessed.
Time Frame: 10 minutes and 30 minutes after injection
Measure: Number; unit: Percentage of Participants
Arm/Group | Current Formulation Adalimumab | New Formulation of Adalimumab
Number analyzed (Participants) | 62 | 62
Percentage of Participants
  10 minutes | 91.9 | 96.8
  30 minutes | 98.4 | 98.4

4. Secondary Outcome: Percentage of Participants With no Erythema in the Draize Scale
Description: Erythema (redness) was assessed.
Time Frame: 10 minutes and 30 minutes after injection
Measure: Number; unit: Percentage of Participants
Arm/Group | Current Formulation Adalimumab | New Formulation of Adalimumab
Number analyzed (Participants) | 62 | 62
Percentage of Participants
  10 minutes | 69.4 | 64.5
  30 minutes | 75.8 | 72.6

5. Secondary Outcome: Percentage of Participants With no Edema in the Draize Scale
Description: Edema (swelling) was assessed.
Time Frame: 10 minutes and 30 minutes after injection
Measure: Number; unit: Percentage of Participants
Arm/Group | Current Formulation Adalimumab | New Formulation of Adalimumab
Number analyzed (Participants) | 62 | 62
Percentage of Participants
  10 minutes | 80.6 | 83.9
  30 minutes | 85.5 | 85.5

6. Secondary Outcome: Percentage of Participants With no Pruritus in the Draize Scale
Description: Pruritus (itching) was assessed.
Time Frame: 10 minutes and 30 minutes after injection
Measure: Number; unit: Percentage of Participants
Arm/Group | Current Formulation Adalimumab | New Formulation of Adalimumab
Number analyzed (Participants) | 62 | 62
Percentage of Participants
  10 minutes | 100 | 98.4
  30 minutes | 98.4 | 98.4

7. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and which did not necessarily have a causal relationship with this treatment.
Time Frame: Adverse events were collected from the time of study drug administration until 70 days following discontinuation of study drug. Serious Adverse Events were collected from the time the participant signed the informed consent.
Measure: Number; unit: participants
Arm/Group | Current Formulation Adalimumab | New Formulation of Adalimumab
Number analyzed (Participants) | 63 | 62
participants | 2 | 1

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of study drug administration until 70 days following discontinuation of study drug. In addition, SAEs were collected from the time the participant signed the study-specific informed consent.
Arm/Group | Current Formulation Adalimumab | New Formulation of Adalimumab
Serious Adverse Events (participants affected / at risk) | 0/63 | 0/62
Other Adverse Events (participants affected / at risk) | 2/63 | 1/62
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Current Formulation Adalimumab (N=63) | New Formulation of Adalimumab (N=62)
PHARYNGITIS (Infections and infestations) | 1 | 0
PROTEIN URINE PRESENT (Investigations) | 0 | 1
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.